CLINICAL TRIAL: NCT02508558
Title: Validation of Methods for Evaluating Operation Force, Motion and Visual Perception in Weightlessness
Acronym: HopMot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-102
Record Dates: First submitted 2015-07-21; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Measurements under different gravity states (Other): motion perception and locomotor operation performance under different gravity states
  Interventions: Other: motion perception and locomotor operation performance measurements; Other: parabolic flight

INTERVENTIONS:
Other: motion perception and locomotor operation performance measurements
Other: parabolic flight

SUMMARY:
Previous studies have neglected two important aspects for the China National Space Administration. First, while biomechanical models are very sensitive to the characteristics of the subjects, data have been collected on subjects with biomechanical characteristics very different from those of "typical" Chinese astronauts. Second, pure video analysis techniques and kinematic data lack the necessary acceleration information important to understanding the forces exerted during movement and control of human motion. While some studies used force and moment sensors to aid in robot torque control and human joint work estimation, investigators are unaware of any studies performed in a microgravity environment that have combined the kinetic force and moment information with acceleration measurements to enable more reliable motion tracking without the need for acceleration estimation.

This is why MICR0-G sensors and accompanying kinematic video system have been developed in order to provide for detailed analyses of the astronaut movement control strategy (joint forces and torques, kinetic and acceleration measurements). Knowledge of the joint torques permits us to calculate the joint and musculoskeletal dynamics required to execute the microgravity motions, as well to provide insight into the altered movement strategies in reduced gravity as compared to 1-G locomotion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese volunteers (men or women)
* Living in France and affiliated to a French Social Security system
* Aged from 22 to 45
* Body Mass Index from 19 to 25
* Who accepted to take part in the study
* Who has given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
motion perception performance under different gravity states | baseline
  MICR0-G sensors and accompanying kinematic video system analyses of the astronaut movement control strategy (joint forces and torques, kinetic and acceleration measurements).
locomotor operation performance under different gravity states | baseline
  MICR0-G sensors and accompanying kinematic video system analyses of the astronaut movement control strategy (joint forces and torques, kinetic and acceleration measurements).

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France